CLINICAL TRIAL: NCT05626803
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Single Dose, Dose-ranging Study to Determine the Safety and Immunogenicity of Bivalent GI.1 and GII.4 Vaccine Administered Orally to Healthy Volunteers Aged Greater Than or Equal to 18 Years and Less Than or Equal to 80 Years Old.
Brief Title: A Study to Determine the Safety and Immunogenicity of Bivalent GI.1 and GII.4 Vaccines in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA-NVV-202
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Norovirus Infections
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Open Label Sentinel (Experimental): Bivalent GII.4/GI.1 vaccine Bivalent GII.4/GI.1 high dose vaccine (VXA-GII.4-NS plus VXA-G1.1-NN) 1×10 to the power 11 tablets total dose is 2×10 to the power 11 IU/dose (sentinel n=10)
  Interventions: Drug: Open label Bivalent GII.4/GI.1 high dose vaccine 2×10 to the power 11 IU/dose
- Medium Dose Arm (Experimental): Bivalent GII.4/GI.1 vaccine Bivalent GII.4/GI.1 medium dose vaccine (VXA-GII.4-NS plus VXA-G1.1-NN) 5×10 to the power 10 tablets total dose is 1×10 to the power 11 IU/dose (N=50)
  Interventions: Drug: Bivalent GII.4/GI.1 medium dose vaccine 1×10 to the power 11 IU/dose
- High Dose Arm (Experimental): Bivalent GII.4/GI.1 vaccine Bivalent GII.4/GI.1 high dose vaccine (VXA-GII.4-NS plus VXA-G1.1-NN) 1×10 to the power 11 tablets total dose is 2×10 to the power 11 IU/dose (N=50)
  Interventions: Drug: Bivalent GII.4/GI.1 high dose vaccine 2×10 to the power 11 IU/dose
- Placebo Arm (Placebo Comparator): Placebo tablets (N= 25)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Open label Bivalent GII.4/GI.1 high dose vaccine 2×10 to the power 11 IU/dose — The first 10 sentinel subjects will receive open label high dose of active vaccine. Bivalent GII.4/GI.1 high dose vaccine (VXA-GII.4-NS plus VXA-G1.1-NN) 1×10 to the power 11 tablets; total dose is 2×10 to the power 11 IU/dose
  Arms: Open Label Sentinel
Drug: Bivalent GII.4/GI.1 high dose vaccine 2×10 to the power 11 IU/dose — 50 subjects will receive high dose of active vaccine. Bivalent GII.4/GI.1 high dose vaccine (VXA-GII.4-NS plus VXA-G1.1-NN) 1×10 to the power 11 tablets; total dose is 2×10 to the power 11 IU/dose
  Arms: High Dose Arm
Drug: Bivalent GII.4/GI.1 medium dose vaccine 1×10 to the power 11 IU/dose — 50 subjects will receive Bivalent GII.4/GI.1 medium dose vaccine (VXA-GII.4-NS plus VXA-G1.1-NN) 5×10 to the power 10 tablets; total dose is 1×10 to the power 11 IU/dose
  Arms: Medium Dose Arm
Drug: Placebo — 25 subjects will receive matching placebo
  Arms: Placebo Arm

SUMMARY:
This study is designed to evaluate the safety and immunogenicity of two monovalent Norovirus (NoV) oral tableted vaccine candidates, VXA-G1.1-NN and VXA-GII.4-NS co-administered (bivalent delivery) against a matching placebo arm. Bivalent GI.1 and GII.4 vaccines are being investigated for the prevention of noroviral gastroenteritis caused by norovirus GI.1 and GII.4.

DETAILED DESCRIPTION:
Norovirus infections are a leading cause of sporadic and epidemic gastroenteritis across all age groups worldwide. This study is designed as a standard double-blind placebo-controlled single administration, dose ranging study to evaluate the safety and immunogenicity of 2 different doses of VXA-GII.4-NS plus VXA-G1.1-NN (high and medium dose administered orally for the prevention of Norovirus infection), compared with a placebo.

This study will enroll a total of 135 subjects with10 sentinel subjects in an open label period (dosing staggered to not-more-than 2 subjects per 24 hours) and randomize 125 subjects in three arms.

The first 10 sentinel subjects will receive the open label high dose of active vaccine. If no dose-related toxicities are observed, and upon the recommendation of the SMC following review of safety data, subjects will be randomized in a 2:2:1 ratio to one of the 3 study arms to receive active vaccine or placebo. After vaccination on Day 1, the study will include an Active Study Period that runs through 4 weeks after administration (Day 29), and a Follow-up Period of one year for safety and duration of immune response.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for this study, subjects must meet all the following:

1. In stable and good general health, without significant medical illness, based on medical history, physical examination, and vital signs at screening based on investigator judgement.
2. Body mass index (BMI) between >/= 17.0 and </= 35.0 kg/m2 at screening SNG.
3. Available for all planned visits and tele-health appointment, and willing to complete all protocol-defined procedures and assessments (including ability and willingness to swallow multiple small enteric-coated tablets per study dose).
4. Female subjects must not be breastfeeding and must provide a negative pregnancy test at screening and pre-dose.
5. Female subjects must fulfill one of the following criteria:

   i. At least 1 year post-menopausal (defined as amenorrhea for greater than or equal to 12 consecutive months prior to screening without alternative medical cause) or surgically sterile.

   ii. Female subjects of childbearing potential must be willing to use a highly effective form of contraception for 30 days prior to initial vaccination and until 60 days after last vaccination. Acceptable forms are oral, implantable, intrauterine, transdermal, intravaginal, injectable, double barrier or abstinence (subjects using diaphragms must also use condom). The form of contraception must be approved by the investigator.

   iii. Male subjects must agree to practice abstinence from heterosexual intercourse or to use an effective method of birth control as noted above from first vaccination to 60 days after last vaccination. Male subjects must agree to refrain from donating sperm and practice abstinence from all intercourse or to use an effective method of double barrier birth control or condom as noted above from first vaccination to 60 days after last vaccination.
6. Capable of understanding and giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

Key Exclusion Criteria:

The subjects must be excluded from participating in the study if they meet any of the following:

1. Known clotting/bleeding issues and/or personal and family history with increased risk of bleeding or clotting.
2. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months prior to screening and reconfirmed at baseline.
3. Cancer, or treatment for cancer or any procedure or preventive medication for cancer or to prevent recurrence, within past 3 years (excluding fully treated and resolved basal cell carcinoma or squamous cell carcinoma)
4. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus- type 1 and 2
5. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine. Such conditions may include but are not limited to:

   a. Any history of: i. GI malignancy ii. malabsorption iii. pancreatobiliary disorders iv. inflammatory bowel disease v. irritable bowel disease vi. hiatal hernia vii. surgical resection b. History of diagnosis or treatment in past 5 years of: i. esophageal or gastric motility disorder ii. gastro esophageal reflux disorder iii. peptic ulcer iv. cholecystectomy
6. History of any form of angioedema
7. History of serious reactions to vaccination such as anaphylaxis, respiratory problems, hives or abdominal pain
8. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic.
9. Any condition that resulted in the absence or removal of the spleen
10. Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness (as determined by the investigator through medical history and physical exam). (Assessment may be repeated once during Screening Period)
11. Presence of a fever greater than or equal to 38°C measured orally at baseline.
12. Any significant hospitalization within the last year which in the opinion of the investigator or sponsor could interfere with study participation.
13. Any history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

    1. Family or personal history of bleeding or thrombosis.
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments.
    3. History of autoimmune or inflammatory disease.
    4. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to screening:

    i. Recent surgery other than removal/biopsy of cutaneous lesions ii. Immobility (confined to bed or wheelchair for 3 or more successive days) iii. Head trauma with loss of consciousness or documented brain injury iv. Receipt of anticoagulants for prophylaxis of thrombosis v. Recent clinically significant infection, including hospitalization for COVID-19 infection.
14. Any other condition that in the clinical judgement of the investigator would jeopardize the safety or rights of a subject taking the study drug, would render the subject unable to comply within the protocol or would interfere with the evaluation of the study endpoints diagnostic assessments.
15. Positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV) tests at the screening visit.
16. History of GI bleeding including hematochezia (blood in stool) or melena (black stool)
17. Positive urine drug screen for drugs of abuse at screening (positive test for marijuana is not exclusionary; however concurrent use of marijuana during the study Active period through Day 29 is prohibited).
18. Positive breath or urine alcohol test at screening and baseline.
19. Receipt of a licensed vaccine (including any COVID-19 vaccines under emergency use authorization) within 14 days prior to baseline vaccination or planned administration during the study active period (Day 29).
20. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 7 days prior to study drug administration or planned use during the active study period (Day 29).
21. Use of medications known to affect the immune function (e.g., including but not limited to systemic corticosteroids, leukotriene modifiers, and JAK inhibitors) within 2 weeks before study drug administration or planned use during the active study period (Day 29).
22. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study drug administration or planned use during the active study period (Day 29). Low dose daily ASA less than or equal to 100 mg for cardio-protection is not exclusionary.
23. Administration of any investigational vaccine, drug or device within 8 weeks preceding study drug administration, or planned use within the duration of the study
24. Previous participation in a Vaxart Clinical Trial or other NoV vaccine trial unless confirmed receipt of placebo.
25. Donation or use of blood or blood products within 30 days prior to study drug administration or planned donation during the active study period (Day 29).
26. History of drug, alcohol, or chemical abuse within 1 year of screening.
27. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to fish gelatin allergy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Director — Vaxart, Inc.
Locations (3):
- United States (3):
  - Ark Clinical Research, Long Beach, California
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Nucleus Network Pty Ltd, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 135 participants were enrolled between January 2023 and October 2023 in the Unites States.
Groups:
- Bivalent GI.1/GII.4 Vaccine Medium Dose: Participants received a single dose of bivalent GI.1/GII.4 (VXA-G1.1-NN plus VXA-GII.4-NS) medium dose vaccine 5×10^10 tablets. Total dose was 1×10^11 IU/dose.
- Bivalent GI.1/GII.4 Vaccine High Dose: Participants received a single dose of bivalent GI.1/GII.4 (VXA-G1.1-NN plus VXA-GII.4-NS) high dose vaccine 1×10^11 tablets. Total dose was 2×10^11 IU/dose.
- Sentinels Open Label High Dose: Participants received a single dose of open label bivalent GI.1/GII.4 (VXA-G1.1-NN plus VXA-GII.4-NS) high dose vaccine 1×10^11 tablets. Total dose was 2×10^11 IU/dose.
- Placebo: Participants received matching placebo.
Period: Overall Study
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Started | 50 | 50 | 10 | 25
Completed | 50 | 49 | 10 | 25
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): All randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the treatment (vaccine) they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 10 | 25 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 47 | 10 | 25 | 126
  >=65 years | 6 | 3 | 0 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 5 | 11 | 60
  Male | 26 | 30 | 5 | 14 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 2 | 4 | 15
  Not Hispanic or Latino | 42 | 48 | 8 | 21 | 119
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 6 | 3 | 1 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 10 | 11 | 1 | 3 | 25
  White | 32 | 34 | 7 | 17 | 90
  More than one race | 2 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Symptoms of Reactogenicity (Gastrointestinal [GI] and Systemic)
Description: Solicited adverse events (AEs) are predefined signs and symptoms of reactogenicity for which the participants were specifically questioned, and which were noted by the participant in their Solicited Symptom Diary for 7 days after drug administration, including:
  * fever (any temperature 100.4°F or higher)
  * headache
  * myalgia (muscle pain)
  * abdominal pain
  * anorexia (defined as not eating)
  * nausea
  * vomiting
  * diarrhoea
  * malaise/fatigue.
  The severity of each solicited symptoms of reactogenicity was graded by the participant as mild, moderate, severe or life-threatening. Participants with multiple Solicited AEs were only counted once in summarizing overall percentages of Solicited AEs, the highest severity of which was used.
Time Frame: Up to Day 8
Population: SAF: All randomized participants received at least 1 dose of the study drug. Participants were analyzed according to the treatment (vaccine) they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 10 | 25
Participants
  Mild | 20 | 20 | 2 | 9
  Moderate | 3 | 9 | 1 | 5
  Severe | 0 | 0 | 0 | 0
  Life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: Treatment emergent AEs (TEAEs) are defined as AEs that occurred following the first administration of study medication. An unsolicited AE is an observed AE that did not fulfill the conditions prelisted in terms of diagnosis and/or onset window post-vaccination.
  The severity of each AE was graded by the participant as mild, moderate or severe/ life-threatening.
Time Frame: Up to Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 10 | 25
Participants
  Mild | 5 | 9 | 2 | 3
  Moderate | 3 | 1 | 0 | 1
  Severe/ Life-threatening | 0 | 0 | 0 | 1

3. Primary Outcome: Serum - Anti-Vaccine Protein 1 (VP1) GI.1 Immunoglobulin A (IgA) Levels by Meso Scale Discovery (MSD) Assay
Description: Serum levels of Anti-VP1 GI.1 IgA were evaluated using cellular and humoral immune (HI) function assays from blood and mucosal (saliva and nasal swab) samples. 95% confidence intervals were estimated by Clopper-Pearson exact method. Assay is measured in AU/mL.
Time Frame: Day 1 and Day 29
Population: Immunogenicity Analysis Set (IS): All randomized participants who received at least 1 dose of the study drug and had at least one valid immunogenicity result after Day 1. Participants were analyzed according to the treatment (vaccine) they actually received.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
AU/mL
  Day 1 | 461471.1 [294526.0 to 723045.2] | 519763.7 [318805.2 to 847396.3] | 149810.3 [47236.2 to 475125.2] | 533470.9 [255503.2 to 1113846.0]
  Day 29 | 1456125.4 [956707.8 to 2216247.4] | 1913341.7 [1257483.5 to 2911272.0] | 657853.4 [248820.3 to 1739291.7] | 545855.7 [259791.3 to 1146914.6]

4. Primary Outcome: Fold Rise in Serum - Anti-VP1 GI.1 IgA Levels by MSD Assay
Description: Serum levels of Anti-VP1 GI.1 IgA were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. The fold rise was calculated per participant by dividing the antibody concentration (original scale) on Day 29 with antibody concentration at baseline (Day 1). 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: IS: All randomized participants who received at least 1 dose of the study drug and had at least one valid immunogenicity result after Day 1. Participants were analyzed according to the treatment (vaccine) they actually received.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Fold Rise | 3.16 [2.35 to 4.24] | 3.68 [2.80 to 4.84] | 4.39 [2.22 to 8.68] | 1.02 [0.95 to 1.10]
Statistical Analysis 1: Comparison: Bivalent GI.1/GII.4 Vaccine Medium Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; Computed by using ANCOVA model with log transformed data as response variable and treatment as a fixed factor and baseline value as covariate
Statistical Analysis 2: Comparison: Bivalent GI.1/GII.4 Vaccine High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sentinels Open Label High Dose vs Placebo; Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 4, analysis 1]

5. Primary Outcome: Serum - Anti-VP1 GII.4 IgGA Levels by MSD Assay
Description: Serum levels of Anti-VP1 GII.4 IgA were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. 95% confidence intervals were estimated by Clopper-Pearson exact method. Assay is measured in AU/mL.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
AU/mL
  Day 1 | 161875.6 [94846.4 to 276275.2] | 259428.2 [161931.1 to 415627.3] | 210263.7 [59975.1 to 737152.9] | 154353.5 [67958.7 to 350580.5]
  Day 29 | 660009.0 [417023.3 to 1044574.4] | 1132279.0 [789453.9 to 1623977.9] | 1213636.4 [616105.1 to 2390685.1] | 185430.7 [81633.1 to 421208.4]

6. Primary Outcome: Fold Rise in Serum - Anti-VP1 GII.4 IgA Levels by MSD Assay
Description: Serum levels of Anti-VP1 GII.4 IgA were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. The fold rise was calculated per participant by dividing the antibody concentration (original scale) on Day 29 with antibody concentration at baseline (Day 1). 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Fold Rise | 4.07 [2.78 to 5.98] | 4.36 [3.25 to 5.85] | 5.78 [1.82 to 18.33] | 1.20 [0.82 to 1.75]
Statistical Analysis 1: Comparison: Bivalent GI.1/GII.4 Vaccine Medium Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Bivalent GI.1/GII.4 Vaccine High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sentinels Open Label High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]

7. Primary Outcome: Serum - Anti-VP1 GI.1 Immunoglobulin G (IgG) Levels by MSD Assay
Description: Serum levels of Anti-VP1 GI.1 IgG were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. 95% confidence intervals were estimated by Clopper-Pearson exact method. Assay is measured in AU/mL.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
AU/mL
  Day 1 | 581088.4 [375777.2 to 898574.5] | 413505.3 [271032.1 to 630872.5] | 227560.5 [77474.5 to 668397.0] | 585351.0 [324390.2 to 1056245.7]
  Day 29 | 1612583.2 [1089047.2 to 2387797.7] | 1203384.0 [810726.2 to 1786216.9] | 670462.8 [225913.2 to 1989792.5] | 575375.0 [315269.9 to 1050073.1]

8. Primary Outcome: Fold Rise in Serum - Anti-VP1 GI.1 IgG Levels by MSD Assay
Description: Serum levels of Anti-VP1 GI.1 IgG were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. The fold rise was calculated per participant by dividing the antibody concentration (original scale) on Day 29 with antibody concentration at baseline (Day 1). 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Fold Rise | 2.78 [2.07 to 3.72] | 2.91 [2.29 to 3.71] | 2.95 [2.25 to 3.86] | 0.98 [0.93 to 1.04]
Statistical Analysis 1: Comparison: Bivalent GI.1/GII.4 Vaccine Medium Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Bivalent GI.1/GII.4 Vaccine High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sentinels Open Label High Dose vs Placebo; Test type: Superiority; p = 0.0017, ANCOVA; [statistical method as in outcome 4, analysis 1]

9. Primary Outcome: Serum - Anti-VP1 GII.4 IgG Levels by MSD Assay
Description: Serum levels of Anti-VP1 GII.4 IgG were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. 95% confidence intervals were estimated by Clopper-Pearson exact method. Assay is measured in AU/mL.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
AU/mL
  Day 1 | 271643.8 [187461.8 to 393628.7] | 242957.4 [166040.8 to 355504.8] | 213650.0 [90624.7 to 503685.4] | 252459.1 [145831.9 to 437048.4]
  Day 29 | 800970.2 [583219.1 to 1100021.2] | 837784.5 [594378.9 to 1180867.6] | 841249.4 [402948.8 to 1756303.8] | 247733.5 [142572.8 to 430459.9]

10. Primary Outcome: Fold Rise in Serum - Anti-VP1 GII.4 IgG Levels by MSD Assay
Description: Serum levels of Anti-VP1 GII.4 IgG were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. The fold rise was calculated per participant by dividing the antibody concentration (original scale) on Day 29 with antibody concentration at baseline (Day 1). 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Fold Rise | 2.95 [2.15 to 4.04] | 3.45 [2.70 to 4.40] | 3.94 [2.01 to 7.70] | 0.98 [0.89 to 1.09]
Statistical Analysis 1: Comparison: Bivalent GI.1/GII.4 Vaccine Medium Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Bivalent GI.1/GII.4 Vaccine High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sentinels Open Label High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]

11. Primary Outcome: Serum - Anti-VP1 GI.1 Blocking Antibodies (BT50) Titers by MSD Assay
Description: Serum levels of Anti-VP1 GI.1 BT50 were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Titer
  Day 1 | 41.9 [29.5 to 59.6] | 41.3 [28.0 to 60.9] | 20.3 [10.5 to 39.4] | 40.6 [21.7 to 76.0]
  Day 29 | 71.2 [49.6 to 102.3] | 75.4 [50.5 to 112.5] | 33.0 [13.3 to 82.1] | 42.3 [23.5 to 76.4]

12. Primary Outcome: Fold Rise in Serum - Anti-VP1 GI.1 BT50 Titers by MSD Assay
Description: Serum levels of Anti-VP1 GI.1 BT50 were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. The fold rise was calculated per participant by dividing the antibody concentration (original scale) on Day 29 with antibody concentration at baseline (Day 1).
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Fold Rise | 1.71 [1.29 to 2.27] | 1.82 [1.50 to 2.22] | 1.62 [1.01 to 2.60] | 1.04 [0.89 to 1.23]
Statistical Analysis 1: Comparison: Bivalent GI.1/GII.4 Vaccine Medium Dose vs Placebo; Test type: Superiority; p = 0.0059, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Bivalent GI.1/GII.4 Vaccine High Dose vs Placebo; Test type: Superiority; p = 0.0020, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sentinels Open Label High Dose vs Placebo; Test type: Superiority; p = 0.1899, ANCOVA; [statistical method as in outcome 4, analysis 1]

13. Primary Outcome: Serum - Anti-VP1 GII.4 BT50 Titers by MSD Assay
Description: Serum levels of Anti-VP1 GII.4 BT50 were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Titer
  Day 1 | 42.0 [29.4 to 60.0] | 51.8 [36.6 to 73.4] | 48.3 [23.4 to 99.7] | 38.4 [23.4 to 63.2]
  Day 29 | 108.7 [80.3 to 147.0] | 138.5 [100.9 to 190.0] | 123.1 [64.1 to 236.5] | 40.6 [25.1 to 65.6]

14. Primary Outcome: Fold Rise in Serum - Anti-VP1 GII.4 BT50 Titers by MSD Assay
Description: Serum levels of Anti-VP1 GII.4 BT50 were evaluated using cellular and HI function assays from blood and mucosal (saliva and nasal swab) samples. The fold rise was calculated per participant by dividing the antibody concentration (original scale) on Day 29 with antibody concentration at baseline (Day 1). 95% confidence intervals were estimated by Clopper-Pearson exact method.
Time Frame: Day 1 and Day 29
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
Number analyzed (Participants) | 50 | 49 | 10 | 25
Fold Rise | 2.58 [1.96 to 3.40] | 2.67 [1.95 to 3.65] | 2.55 [1.33 to 4.89] | 1.06 [0.92 to 1.22]
Statistical Analysis 1: Comparison: Bivalent GI.1/GII.4 Vaccine Medium Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Bivalent GI.1/GII.4 Vaccine High Dose vs Placebo; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sentinels Open Label High Dose vs Placebo; Test type: Superiority; p = 0.0020, ANCOVA; [statistical method as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: For TEAEs: Up to Day 29 For SAEs and all-cause mortality: Up to Day 180
Description: For AEs and SAEs, SAF: All randomized participants who received at least 1 dose of the study drug. Participants were analyzed according to the treatment (vaccine) they actually received.
  For all-cause mortality, Full Analysis Set (FAS): All participants who were randomized. The analyses using FAS were based upon the randomization arm allocated. participants were analyzed according to the treatment (vaccine) planned.
Arm/Group | Bivalent GI.1/GII.4 Vaccine Medium Dose | Bivalent GI.1/GII.4 Vaccine High Dose | Sentinels Open Label High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/10 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/10 | 0/25
Other Adverse Events (participants affected / at risk) | 8/50 | 10/50 | 2/10 | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bivalent GI.1/GII.4 Vaccine Medium Dose (N=50) | Bivalent GI.1/GII.4 Vaccine High Dose (N=50) | Sentinels Open Label High Dose (N=10) | Placebo (N=25)
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT05626803/Prot_SAP_000.pdf